CLINICAL TRIAL: NCT01534520
Title: Self-administered Intravaginal 2% Lidocaine Gel Prior to Intrauterine Device Insertion in Nulliparous Women: a Randomized Controlled Trial
Brief Title: Self-administered Intravaginal 2% Lidocaine Gel Prior to Intrauterine Device Insertion in Nulliparous Women
Acronym: LIVIIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Sharon Achilles, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFP-RBR001
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Intrauterine Device; Pain; Lidocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine; K-Y jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Intravaginal 2% lidocaine gel (Experimental): Intravaginal insertion of 4mL of 2% lidocaine gel
  Interventions: Drug: Lidocaine
- Group 2: Intravaginal placebo gel (Placebo Comparator): Intravaginal insertion of 4mL of placebo gel ( K-Y Jelly)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Intravaginal insertion of 4mL 2% lidocaine gel
  Other Names: Lidocaine Jelly; Lidocaine Hydrochloride
  Arms: Group 1: Intravaginal 2% lidocaine gel
Drug: Placebo — KY Jelly
  Other Names: K-Y Jelly; water based lubricant
  Arms: Group 2: Intravaginal placebo gel

SUMMARY:
This study is designed to evaluate if self-inserted intravaginal 2% lidocaine gel is effective at decreasing pain during intrauterine device insertion in nulliparous women.

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are among the most effective forms of reversible contraception. Numerous studies demonstrate their safety and efficacy in nulliparous women, however, uptake of IUDs in this group is low. One of the major barriers to women obtaining IUDs is fear of pain during insertion, as studies do demonstrate that nulliparous women experience more pain than parous women during IUD insertion. Studies evaluating various methods for pain control during IUD insertion have shown conflicting results, leaving the question unanswered as to what is the best method to decrease pain during IUD insertion.

This study aims to evaluate a novel approach to pain control by having women self-insert lidocaine gel into the vagina at least 5 minutes prior to IUD insertion. This will overcome some of the barriers from other studies where there may not have been ample time for the lidocaine to take effect, while at the same time eliminating the need for women to have multiple speculum exams. Although this is a novel approach to administering an anesthetic, we believe women will be interested in any intervention that may potentially alleviate pain during IUD insertion.

If this study does demonstrate that pain is decreased with self-inserted lidocaine compared to placebo gel, this will potentially eliminate one large barrier to nulliparous women receiving IUDs. Increased uptake of highly effective contraception in nulliparous women is just one of the many steps necessary towards decreasing unintended pregnancy.

ELIGIBILITY:
Inclusion criteria:

* Nulliparous, as defined in this study as no history of pregnancy ≥ 24 weeks gestational age
* Desires insertion of either levonorgestrel-releasing IUD (LNG-IUD) or copper T380A IUD (Cu-IUD)
* No history of pregnancy in the last 6 weeks
* Able to provide written informed consent in English and comply with all study procedures

Exclusion criteria:

* Known allergy or hypersensitivity to lidocaine or other amino amide local anesthetics
* Prior failed IUD insertion
* Prior IUD use
* Use of narcotic or benzodiazepine medication within the last 24 hours
* U.S. Centers for Disease Control Medical Eligibility Criteria (MEC) category 3 or 4 classification for use of an IUD
* Positive pregnancy test or reasonable risk of pregnancy due to unprotected heterosexual intercourse since the last menstrual period

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B Rapkin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rapkin RB, Achilles SL, Schwarz EB, Meyn L, Cremer M, Boraas CM, Chen BA. Self-Administered Lidocaine Gel for Intrauterine Device Insertion in Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2016 Sep;128(3):621-8. doi: 10.1097/AOG.0000000000001596. PMID 27500351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 79 women presenting for IUD insertion at OPC, UPP, and GMO were approached for participation.
Pre-assignment Details: * 2 patients were removed from the study. Patients were considered screen failures before randomization to an arm.
  * 18 declined participation; 10 (56%) reported "time concerns" as their primary reason for declining.
Groups:
- Group 1: Intravaginal 2% Lidocaine Gel: 4 ml of 2% lidocaine gel for self vaginal insertion
- Group 2: Intravaginal Placebo Gel: Intravaginal insertion of 4ml of placebo gel (K-Y Jelly)
Period: Overall Study
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel
Started | 30 | 29
Completed | 30 | 28 (1 subject withdrew consent at time of uterine sound attempt due to intolerable pain)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomization is blinded.
Groups:
- Group 1: Intravaginal 2% Lidocaine Gel: 4mL of 2% lidocaine gel for vaginal self-administration
  )
- Group 2: Intravaginal Placebo Gel: 4mL placebo gel (K-Y Jelly) for vaginal self-administration
- Total: Total of all reporting groups
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Customized [Number; unit: participants] — Randomization was blinded.
  participants
    Between 14-50 | 30 | 29 | 59
Gender [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain From Baseline to IUD Insertion
Description: To assess change in pain from baseline to IUD insertion measured on a visual analog scale (VAS) from 0 mm (no pain) to 100 mm (worst pain in patient's life). This pain assessment was prior to (baseline) and at the time of IUD insertion following vaginal self-administration of study gel (either 2% lidocaine gel or placebo gel).
Time Frame: change in pain score from baseline (before IUD insertion) to time of IUD insertion
Measure: Median (Inter-Quartile Range); unit: change in visual analog scale score
Groups:
- Group 1: Intravaginal 2% Lidocaine Gel: Intravaginal insertion of 4mL of 2% lidocaine gel
  Placebo: KY Jelly
- Group 2: Intravaginal Placebo Gel: Intravaginal insertion of 4mL of placebo gel ( K-Y Jelly)
  Lidocaine: Intravaginal insertion of 5mL 2% lidocaine gel
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel
Number analyzed (Participants) | 30 | 29
change in visual analog scale score | 61 [53 to 71] | 68 [58 to 80]

2. Secondary Outcome: To Evaluate Patient Experience of Self-inserting the Intravaginal Study Gel Prior to IUD
Description: Number of participants who rated self-application of study gel as "some what easy" or "very easy" on Likert scale
Time Frame: After inserting the gel but prior to IUD insertion
Measure: Number; unit: participants who found gel easy to use
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel
Number analyzed (Participants) | 30 | 29
participants who found gel easy to use | 29 | 29

3. Secondary Outcome: Percentage of IUDs Considered by Physicians Easy to Insert
Description: The physician who conducted the study visit and IUD insertion was asked about the difficulty/ease in placing the IUD immediately following the procedure and the percentage of IUD insertions considered to be "easy" was calculated for each study group.
Time Frame: Directly after IUD insertion
Population: Participants in each group self-administered the study gel as per instruction followed by insertion of the IUD by the physician 5 to 15 minutes later.
Measure: Number (95% Confidence Interval); unit: percentage of insertions declared easy
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel
Number analyzed (Participants) | 30 | 29
percentage of insertions declared easy | 87 [69 to 96] | 64 [44 to 81]

4. Secondary Outcome: Need for Pain Medication up to 7 Days
Description: Number of women taking pain medication for at least one day following IUD insertion
Time Frame: 7 days post-insertion
Measure: Number; unit: participants
Arm/Group | Group 1: Intravaginal 2% Lidocaine Gel | Group 2: Intravaginal Placebo Gel
Number analyzed (Participants) | 30 | 28
participants | 24 | 27

ADVERSE EVENTS:
Groups:
- Placebo: Intravaginal insertion of 4mL placebo gel
  Placebo: KY Jelly
- Study Drug: Intravaginal insertion of 4mL 2% lidocaine gel
  Lidocaine: Intravaginal insertion of 4mL 2% lidocaine gel
Arm/Group | Placebo | Study Drug
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 1/29 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | Study Drug (N=30)
Intolerable Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Pain at time of IUD insertion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes